CLINICAL TRIAL: NCT03731338
Title: An Exploratory Study of a Nurse-Led Rapid Access Chest Pain Clinic, From the Patients' Perspectives
Brief Title: Nurse-Led Rapid Access Chest Pain Clinic
Status: Completed | Type: Observational
Sponsor: The Royal Wolverhampton Hospitals NHS Trust (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2017CAR95
Record Dates: First submitted 2018-10-29; First posted 2018-11-06 (Actual); Last update posted 2019-10-02 (Actual); Status verified 2019-10

CONDITIONS: Chest Pain
MeSH Terms: conditions — Chest Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Reassured and discharged: patients who are reassured and discharged after first attendance
- Further diagnostic testing: Patients who went on to have further diagnostic testing

SUMMARY:
This study aims to ascertain the lived experiences of 6 patients attending a nurse-led chest pain clinic via an interview, and to understand the demographics of referred patients.

DETAILED DESCRIPTION:
A qualitative analysis of a nurse-led chest pain clinic will be undertaken to improve understanding of patient experience. Patients who have used this service will be invited to take part in an interview. Patients will be split in to two groups: those reassured and discharged after first attendance, and those who went on to have further diagnostic testing. The aim is to interview three patients from each group to compare experiences and perceptions of a service which previously would have been undertaken by physicians, but is now completely nurse-led.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have attended the chest pain clinic in the last four month months
* Eighteen years-of-age and older
* Able to give valid consent
* English speaking

Exclusion Criteria:

* Non-English speaking patients
* Patients under 18 years of age
* Patients with any cognitive impairment.
* Any vulnerable patients (defined by the mental health act 2005 as anyone lacking capacity to make decisions, ie, someone with severe impairment in the functioning of the brain).
* Offenders in the care of prison services (for logistical reasons)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population targeted will be patients referred to the rapid access chest pain clinic undertaken once a week by the researcher or one colleague on alternate weeks.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2017-12-21 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
Explore the lived experiences through interview | 1 hour
  Explore the lived experiences of patients attending a nurse-led rapid access chest pain clinic through interview of participants

SECONDARY OUTCOMES:
Outcome of the consultation Effects through interview | 1 hour
  Understand if these experiences are affected in any way by the outcome of the consultation through interview of participants

CONTACTS AND LOCATIONS:
Overall Officials: Justin Lewis, Principal Investigator — The Royal Wolverhampton NHS Trust
Locations (1):
- New Cross Hospital, Wolverhampton, West Midlands, United Kingdom